CLINICAL TRIAL: NCT06705790
Title: Exploring the Feasibility and Urogenital Benefits of Pelvic Floor Muscle Training in Individuals with Motor-incomplete Spinal Cord Injury
Brief Title: Exploring the Benefits of Pelvic Floor Muscle Training on Bladder, Bowel, and Sexual Function in People with Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Tania Lam, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H21-02281; PTJ-166040 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2024-11-18; First posted 2024-11-26 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injury; Pelvic Floor Muscle Training; Bladder; Bowel; Sexual Health
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pelvic Floor Muscle Training Group (Experimental)
  Interventions: Behavioral: Pelvic Floor Muscle Training

INTERVENTIONS:
Behavioral: Pelvic Floor Muscle Training — Pelvic floor muscle training 5x/week for 12-weeks

SUMMARY:
The goal of this trial is to learn about the feasibility and benefits of delivering a pelvic floor muscle training program to people with motor-incomplete spinal cord injury. The main questions it aims to answer are:

1. To evaluate the feasibility of delivering a pelvic floor muscle training program to people with spinal cord injury. The investigators will examine recruitment rate, compliance and adherence to the intervention and other study protocols, adverse events, and participant perspectives of the study protocols.
2. To explore the potential effectiveness of pelvic floor muscle training on pelvic floor, bladder, bowel, and sexual function.

Participants will be asked to complete a pelvic floor muscle training program for 3 months. At the beginning, middle, and end of the program, researchers will conduct a series of tests to determine the feasibility and potential effectiveness of this program.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 19 years of age.
* Have a non-progressive, motor-incomplete spinal cord injury that is at or above the T12 neurological level at least 12 months ago.
* Have symptoms of bladder, bowel, and/or sexual dysfunction that are caused by your spinal cord injury.
* Have stable management of spinal cord related secondary health concerns (e.g., spasticity, neuropathic pain).
* Are able to speak and understand English.

Exclusion Criteria:

* Are currently pregnant, have been pregnant within the past 6 months, or are planning to become pregnant in the next 6 months.
* Have had urogenital surgery within the past 12 months.
* Have received Botox bladder injections within the past 4 weeks, or anticipate receiving an injection in the next 6 months.
* Have presence of severe medical issue that in the investigator's judgement would adversely affect the participant's participation in the study. Examples include, but are not limited to pressure sores, cardiovascular disease, and unmanaged diabetes.
* Have any permanent metal fixtures in their head (excluding dental fillings), or pacemakers, stimulators, or implanted medication pumps.
* Have a history of seizures, are taking medications that lower the seizure threshold, or experience recurring headaches.
* Have a condition for which exercise is contraindicated.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Recruitment Rate | Through study completion, up to 12 weeks
  Recruitment rate will be evaluated by number of participants approached, screened for eligibility, as well as reasons for exclusions.
Feasibility - Compliance | Through study completion, up to 12 weeks
  Compliance will be tracked by the adherence of participants to the prescribed exercise program, with reasons for missed sessions or drop-outs noted.
Feasibility - Adverse Events | Through study completion, up to 12 weeks
  Any adverse events to study protocols will be recorded.
Feasibility - Acceptability | Through study completion, up to 12 weeks
  The acceptability of the intervention will be evaluated using a 7-point Likert scale to rate participants' enjoyment of the exercise program and whether they felt the program was beneficial for improving their bladder, bowel, and/or sexual function.

SECONDARY OUTCOMES:
Incontinence Quality of Life Questionnaire (I-QoL) | From enrollment to within 2 weeks of completing the study intervention
  Participants will be asked to respond to 22 questions about how urinary incontinence impacts their quality of life using a 5-point scale with values ranging from 1 (extremely) to 5 (not at all). The questionnaire probes three subdomains of how incontinence may affect quality of life: avoidance and limiting behavior, psychosocial impact, and social embarrassment.
Neurogenic Bladder Symptoms Score (NBSS) | From enrollment to within 2 weeks of completing the study intervention
  Participants will be asked to respond to 24 questions regarding the severity of their bladder symptoms secondary to neurological injury. Questions cover three subdomains: incontinence, storage and voiding, and consequences.
3-Day Bladder Diary | From enrollment to within 2 weeks of completing the study intervention
  Participants will be asked to record information regarding their fluid intake (i.e., time, volume, and type) and voids (i.e., time, volume, leaks, and pad change) for three days. The investigators will use the combined information on intake and voids to make a clinical summary of the participants urinary function.
Timed Bowel Movement | From enrollment to within 2 weeks of completing the study intervention
  Participants will be asked to how long their bowel movements take, and what (if any) aids they used to complete the bowel movement (e.g. suppository, laxatives, digital stimulation/evacuation, etc).
Neurogenic Bowel Dysfunction Score (NBDS) | From enrollment to within 2 weeks of completing the study intervention
  Participants will be asked to complete the NBDS which asks 11 questions to clinically assess the severity of their bowel dysfunction symptoms. Results of this questionnaire provide a score from 0 to 47, where a higher score represents more severe bowel symptoms.
International Index of Erectile Function (IIEF) Questionnaire (Males only) | From enrollment to within 2 weeks of completing the study intervention
  Male participants will be asked to complete the IIEF questionnaire which askes 15 questions to clinically assess sexual health in 5 domains: erectile function (possible score of 0-30), orgasmic function (possible score of 0-10), sexual desire (possible score of 0-10), intercourse satisfaction (possible score of 0-15), overall satisfaction (possible score of 0-10). In all domains, a higher score represents more severe sexual dysfunction.
Female Sexual Function Index (FSFI) Questionnaire (Females Only) | From enrollment to within 2 weeks of completing the study intervention
  Female participants will be asked to complete the FSFI questionnaire which askes 19 questions to clinically assess sexual health in 6 domains: desire (possible score of 1.2-6), arousal (possible score of 0-6), lubrication (possible score of 0-6), orgasm (possible score of 0-6), satisfaction (possible score of 0.8-6), and pain (possible score of 0-6). In all domains, a higher score represents a less sexual dysfunction.
Sexual Quality of Life Questionnaire - Male/Female | From enrollment to within 2 weeks of completing the study intervention
  Male and female participants will both be asked to complete their sex-specific version of this questionnaire. This questionnaire asks respondents to rate 11 statements (male, possible score of 11-66) or 18 statements (female, possible score of 18-108) according to how much they agree or disagree with it. For both the male and female version of the questionnaire, a higher score represents better sexual quality of life.
Pelvic Floor Electromyography | From enrollment to within 2 weeks of completing the study intervention
  PFM function (i.e., endurance and motor control) will be assessed using surface electromyography (EMG). Disposable surface electrodes will be placed perianally to record from the pelvic floor muscles, and other electrodes will be placed over the relevant muscles in the trunk and legs. Participants will be asked to attempt various contractions of their pelvic floor muscles including a maximal, isolated pelvic floor contraction; a sustained pelvic floor contraction to assess endurance; and a rapid contract-relaxation task to assess motor control.
Effectiveness of Cueing | From enrollment to within 2 weeks of completing the study intervention
  Researchers will ask participants about their perceived effectiveness of verbal instructions and feedback strategies used in the pelvic floor muscle training sessions for facilitating voluntary activation of the pelvic floor.
Transcranial Magnetic Stimulation (TMS) Assessment | From enrollment to within 2 weeks of completing the study intervention
  The investigators will assess the connection of the neural pathways between the brain and pelvic floor using transcranial magnetic stimulation (TMS). TMS will be delivered over the primary motor cortex in the brain, and motor evoked potentials (MEPs) will be recorded using surface electromyography from the pelvic floor. Participants will be instruction to maintain a sub-maximal contraction of the pelvic floor during the experiment, while TMS pulses are delivered at a variety of intensities.
Pudendal Somatosensory Evoked Potential (SEP) Assessment | From enrollment to within 2 weeks of completing the study intervention
  Pudendal nerve function will be assessed through an somatosensory evoked potential (SEP) assessment. Non-painful electrical stimulations of up to 1ms in duration will be delivered to the pudendal nerve via the electrodes placed over the genitals while the investigators simultaneously use an electroencephalography (EEG) cap to record from the somatosensory cortex.
Transperineal Ultrasound | From enrollment to within 2 weeks of completing the study intervention
  Pelvic floor muscle function will be assessed through transperineal ultrasound. An ultrasound probe will be placed on the perineum to visualize the pelvic floor and other relevant pelvic structures (e.g. bladder, urethra, vaginal canal, sphincters, pelvic bones). Ultrasound images and recordings will be taken while the participant is at rest and as they attempt PFM contractions.

CONTACTS AND LOCATIONS:
Overall Officials: Tania Lam, PhD, PT, Principal Investigator — University of British Columbia, ICORD
Locations (1):
- Blusson Spinal Cord Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No